CLINICAL TRIAL: NCT05192408
Title: Multi-component Intervention for Reducing Fear of Falling in Community-dwelling Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Healthcare Group Polyclinics (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/00742
Record Dates: First submitted 2021-12-30; First posted 2022-01-14 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Fear of Falling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants and study team members who carry out intervention(nurses) will not be masked. Outcome assessors will be study team members from different clinics as participants or study team members who were not involved in intervention, and will thus be unaware of participants' allocated group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-component intervention (Experimental): Individual intervention will comprise:
  1. Cognitive- behavioral therapy (CBT) which includes: - Behavioural activation, cognitive restructuring, promotion of safety, relaxation techniques
  2. Exercise recommendation utilizing current Exercise in older adults Patient Education Materials (PEMs) and videos, tailored based on frailty level and readiness to progress - Components include balance and strength
  3. Use of motivational interviewing (MI) techniques for goal setting
  There will be 4 sessions in total. Initial sessions will be carried out face to face or via videoconferencing platform if participant prefers due to ongoing COVID-19 pandemic. Subsequent sessions will be carried out via telephone.
  Initial sessions will last around 30 minutes and subsequent sessions will last 15 to 30 minutes.
  Interventions: Behavioral: Multi-component intervention
- Usual Care (Other): Patient Education Materials (PEMs) on:
  1. Exercise in older adults (Stay Active, Stay Strong and Stay Steady) - 3 different levels tailored to frailty level and for progression
  2. Falls prevention
  3. FoF
  Interventions: Other: Usual Care

INTERVENTIONS:
Behavioral: Multi-component intervention — Individual intervention will comprise:
  1. Cognitive- behavioral therapy (CBT) which includes: - Behavioural activation, cognitive restructuring, promotion of safety, relaxation techniques
  2. Exercise recommendation utilizing current Exercise in older adults Patient Education Materials (PEMs) and videos, tailored based on frailty level and readiness to progress - Components include balance and strength
  3. Use of motivational interviewing (MI) techniques for goal setting
  There will be 4 sessions in total. Initial sessions will be carried out face to face or via videoconferencing platform if participant prefers due to ongoing COVID-19 pandemic. Subsequent sessions will be carried out via telephone.
  Arms: Multi-component intervention
Other: Usual Care — Patient Education Materials
  Arms: Usual Care

SUMMARY:
In the short term, the study will provide insight into the effectiveness of multi-component intervention for reducing Fear of falling (FoF) in community-dwelling older adults. Effective interventions will be incorporated into existing programs for frailty and falls prevention in primary care. Reducing FoF will break the cycle of physical activity restriction, functional decline and further falls in older adults. Long term potential benefits include improving the health status of older adults and thus reducing healthcare utilization.

The primary aim is to compare the effectiveness of a multi-component intervention comprising exercise recommendations, cognitive behavioural therapy (CBT) components and motivational interviewing (MI) based telephone review against usual care for reducing Fear of Falling (FoF) in community- dwelling older adults.

Secondary aims include to compare the effectiveness of the multi-component intervention against usual care for increasing physical activity and reducing falls in community- dwelling older adults.

The hypothesis is that the multi-component intervention will be more effective as compared to usual care for reducing FoF and falls and increasing physical activity in community- dwelling older adults.

DETAILED DESCRIPTION:
In the short term, the study will provide insight into the effectiveness of multi-component intervention for reducing Fear of falling (FoF) in community-dwelling older adults. Effective interventions will be incorporated into existing programs for frailty and falls prevention in primary care. Reducing FoF will break the cycle of physical activity restriction, functional decline and further falls in older adults. Long term potential benefits include improving the health status of older adults and thus reducing healthcare utilization.

The primary aim is to compare the effectiveness of a multi-component intervention comprising exercise recommendations, cognitive behavioural therapy (CBT) components and motivational interviewing (MI) based telephone review against usual care for reducing Fear of Falling (FoF) in community- dwelling older adults.

Secondary aims include to compare the effectiveness of the multi-component intervention against usual care for increasing physical activity and reducing falls in community- dwelling older adults.

The hypothesis is that the multi-component intervention will be more effective as compared to usual care for reducing FoF and falls and increasing physical activity in community- dwelling older adults.

Sample size was calculated with reference to effect sizes from meta-analyses where effect sizes of 0.28 and 0.33 were found.

The sample size calculation was based on effect size of 0.3 difference in FoF between the intervention and comparator groups; with power of 80% and significance level of 0.05, 175 patients will be needed in each group. Assuming attrition rate of 20%, 210 participants in each group, or a total of 420 participants, would be needed.

Recruitment procedures Recruitment will take place at all National Healthcare Group Polyclinics over a period of 12 months.

All healthcare staff including doctors, nurses, physiotherapists and care coordinators (CCs) in recruiting clinics will be briefed about the study and inclusion and exclusion criteria. Potential participants will be recruited on a case encounter basis when they attend at the clinics for follow-up visits. The above-mentioned healthcare staff will refer potential participants who meet the inclusion criteria to any of the study team members. Study team members who encounter suitable potential participants will refer them to another study team member in clinic for recruitment if available, i.e., nurses in study team may cross refer their patients to each other for recruitment.

Study team members proficient in potential participants' language will explain the study and clarify any doubts using the Participant Information Sheet, take written informed consent and administer the baseline questionnaire.

Data Collection Tools III) Fear of falling (FoF) will be screened using the Single Question on FoF and Activity Restriction (SQ-FAR) and measured using the Short Falls Efficacy Scale - International (FES-I) The SQ-FAR is a single question 'Are you afraid of falling?' used as a screening tool for FoF. It was found to have moderate agreement of 87.8% (Kappa=0.57) with the Falls Efficacy Scale-International (FES-I) in community dwelling adults aged 65 to 70 years old. Responses include 'no', 'yes' and 'yes, a lot', 'yes' and 'yes, a lot' indicate presence of FoF.

The Short FES-I is a 7-item measure of "fear of falling" and has been demonstrated to have good reliability and validity. It was also evaluated in Malaysia and showed good internal consistency, test-retest reliability, construct validity, and responsiveness, with Cronbach's alpha of 0.905 and intraclass correlation coefficient 0.997 for the English version. Scores are calculated by totaling responses for each item, with a range from minimum 7 (no concern about falling) to maximum 28 (severe concern about falling). 7 to 8 points indicates low concern, 9 to 13 indicates moderate concern and 14 to 28 indicates high concern.

IV) Physical Activity levels will be measured using the Incidental and Planned Exercise Questionnaire: Weekly Average (IPEQ -WA) The IPEQ consists of 10 questions which measure type and amount of physical activity and provides estimates of the frequency and duration of planned exercise and day-to-day activities. Validation in a population of older adults showed that IPAQ-WA had excellent test-retest reliability, with intraclass correlation coefficient 0.87 and was able to discriminate differences in physical activity levels between groups differentiated by sex, age and fall risk factors. Total time spent is summed across all components and expressed as hours per week. The score is derived from multiplying frequency score and duration score to create a total duration for the week score.

Statistical and analytical plans Demographic and clinical data, falls, FoF scores and (IPEQ-WA) scores will be reported using descriptive statistics. Paired t-test will be used to compared the differences in FoF scores, number of falls and IPEQ-WA scores pre and post intervention. Independent t-test will be used to compare differences in FoF score, number of falls and IPEQ-WA scores in intervention group and comparator group at 3 months and 6 months post intervention.

Ethical considerations Informed Consent Attending healthcare professionals will refer eligible participants to members of the study team on the day of the clinic visit. Trained study team members proficient in potential participants' language will explain the study and clarify any doubts using the Participant Information Sheet. Participants will be given the information sheet about the research study and informed that they could withdraw from the study anytime. The contact details of the PI and DSRB would be given to them to allow them to raise any queries regarding the study.

Potential participants will be given adequate time to consider before making a decision whether or not to participate. If the individual fulfils the inclusion criteria and agrees for research participation, written consent will be taken.

Confidentiality of Data and Patient Records Hard copy data will be stored in designated locked cabinet(s) or room(s). Electronic data will be stored in a secured computer that is password protected. All hard copy or electronic data will be accessible to authorized study team members only.

ELIGIBILITY:
Inclusion Criteria:

* Older adults aged 65 and above
* Followed up at National Healthcare Group Polyclinics for any chronic condition
* Able to communicate in English, Mandarin, Malay
* Reports Fear of falling as screened by single question

Exclusion Criteria:

* Unable to agree to participation e.g., due to cognitive impairment
* Unable or unsafe to participate in any exercise as determined by clinician e.g., terminal illness, uncontrolled hypertension, immobility
* Unable to participate in telephone sessions e.g., due to hearing impairment
* Known psychiatric condition on treatment

Ages: 65 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Fear of Falling (FoF) | 3 months
  FoF as measured by short FES-I

SECONDARY OUTCOMES:
Number of falls | 3 months
  Number of falls
Physical Activity | 3 months
  Physical Activity as measured by IPEQ-WA

CONTACTS AND LOCATIONS:
Locations (1):
- National Healthcare Group Polyclinics, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Drahota A, Udell JE, Mackenzie H, Pugh MT. Psychological and educational interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2024 Oct 3;10(10):CD013480. doi: 10.1002/14651858.CD013480.pub2. PMID 39360568